CLINICAL TRIAL: NCT02781220
Title: Implications for Management of PET Amyloid Classification Technology in the Imaging Dementia(IDEAS) Trial
Acronym: IMPACT2
Status: Terminated | Type: Observational
Why Stopped: IRB Study Closure - No HRPP Progress Update
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 90351
Record Dates: First submitted 2016-05-18; First posted 2016-05-24 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment; Dementia; Alzheimer's Disease
Keywords: MCI; Dementia; amyloid PET; physician diagnosis; Alzheimer's disease; AD; PET imaging; Appropriate Use Criteria; patient-reported outcomes; patient adherence
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Qualifying participants: All consented IDEAS trial participants will have additional data collected: visual and semi-quantitative software aided amyloid PET scan interpretation, care partner questionnaires and documented provider diagnosis, diagnostic confidence, and management plan following the IMPACT design

SUMMARY:
The main purpose of this study is to build upon the evidence captured in the Imaging Dementia - Evidence for Amyloid Scanning (IDEAS; NCT02420756) trial to include valuable information regarding patient-reported outcomes and physician confidence in diagnosis and management based on the Implications for Management of PET Amyloid Classification Technology (IMPACT; NCT number not yet assigned) trial design.

DETAILED DESCRIPTION:
The primary purpose of this prospective, observational study is to examine the benefit of amyloid positron emission tomography and computed tomography (PET/CT) scan in clinical practice for participants at our site that are enrolled in the IDEAS (NCT02420756) trial. To accomplish this, when a clinician has ordered an amyloid PET scan, the investigators will assess the impact of [18F]Flutemetamol PET/CT scans on 1) physician diagnosis and management as it relates to care practices and drug management, and 2) patient reported outcomes in patients evaluated in the Cognitive Disorders Clinic at the University of Utah and meeting Appropriate Use Criteria (AUC) for clinical amyloid PET/CT scans. A secondary purpose is to compare the semi-quantitative assessment of amyloid plaque burden using vendor supplied software and standard visual assessment of amyloid positivity.

The primary hypothesis is that, in diagnostically uncertain cases, knowledge of amyloid status as determined by amyloid PET/CT scans may alter patient diagnosis and management and lead to significant changes in patient and family reported outcomes. A secondary hypothesis is that vendor supplied semi-quantitative assessment of amyloid plaque positivity will be superior to standard visual criteria assessments.

Objectives

AIM 1: to assess the change in diagnosis and management, related to care practices and drug management of adult patients being evaluated for cognitive deficits and meeting Appropriate Use Criteria (AUC)

AIM 2: to assess the change of amyloid PET/ CT scans on patient-reported outcomes involving care partner confidence and satisfaction

AIM 3: to assess confidence increase through use of vendor supplied semi-quantitative software

AIM 4: to assess adherence to identified patient management related to care practices and drug management

ELIGIBILITY:
Inclusion Criteria:

* 65 and older;
* Medicare beneficiary;
* Diagnosis of mild cognitive impairment (MCI) or dementia, according to Diagnostic and Statistical Manual - IV (DSM-IV) and/or National Institutes of Aging-Alzheimer's Association criteria, verified by a dementia specialist within 24 months (American Psychiatric Association. 2000; McKhann et al. 2011; Albert et al. 2011);
* Meets AUC:
* Cognitive complaint verified by objectively confirmed cognitive impairment;
* The etiologic cause of cognitive impairment is uncertain after a comprehensive evaluation by a dementia specialist, including general medical and neurological examination, mental status testing including standard measures of cognitive impairment, laboratory testing, and structural neuroimaging as below;
* Alzheimer's disease is a diagnostic consideration;
* Knowledge of amyloid PET status is expected to alter diagnosis and management.
* Head MRI and/or CT within 24 months prior to enrollment;
* Clinical laboratory assessment within the 12 months prior to enrollment: complete blood count (CBC), standard blood chemistry profile, thyroid stimulating hormone (TSH); vitamin B12;
* Able to tolerate amyloid PET required by protocol, to be performed at a participating PET facility;
* English or Spanish speaking (for the purposes of informed consent);
* Willing and able to provide consent. Consent may be by proxy.

Exclusion Criteria:

* Normal cognition or subjective complaints that are not verified by cognitive testing.
* Knowledge of amyloid status, in the opinion of the referring dementia expert, may cause significant psychological harm or otherwise negatively impact the patient or family.
* Scan is being ordered solely based on a family history of dementia, presence of apolipoprotein E, or in lieu of genotyping for suspected autosomal mutation carriers.
* Scan being ordered for nonmedical purposes (e.g., legal, insurance coverage, or employment screening).
* Cancer requiring active therapy (excluding non-melanoma skin cancer);
* Hip/pelvic fracture within the 12 months prior to enrollment;
* Body weight exceeds PET scanner weight limit;
* Life expectancy less than 24 months based on medical co-morbidities;
* Residence in a skilled nursing facility.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants must be Medicare beneficiaries referred by qualified dementia specialists and must meet AUC for amyloid PET (Johnson et al. 2013).
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-07; Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Percentage of change in care practices after amyloid PET scan | Visit 1, 30 days prior to scan and Visit 4, 90 days after scan
  % of 13 care practices that differ before and after the amyloid PET scan

SECONDARY OUTCOMES:
Percentage of change in drug management options after amyloid PET | Visit 1, 30 days prior to scan and Visit 4, 90 days after scan
  % of drug management options that differ before and after the amyloid PET scan
Change in % likelihood of Alzheimer's disease (AD) diagnosis after amyloid PET scan | Visit 1, 30 days prior to scan and Visit 4, 90 days after scan
  Difference in % of AD likelihood identified before and after the amyloid PET scan
Percentage of change in leading diagnosis after amyloid PET | Visit 1, 30 days prior to scan and Visit 4, 90 days after scan
  % of leading diagnosis that differ before and after amyloid PET scan
Change in physician confidence in leading diagnosis | Visit 1, 30 days prior to scan and Visit 4, 90 days after scan
  Difference in 5-point scale of physician confidence in leading diagnosis before and after amyloid PET scan
Change in care partner's confidence in diagnosis after amyloid PET | Visit 1, 30 days prior to scan, Visit 4, 90 days after scan, Visit 5, 180 days after scan and Visit 6, 270 days after scan
  Difference in 5-point scale of care partner confidence in diagnosis before and after amyloid PET scan
Change in care partner satisfaction with evaluation after amyloid PET | Visit 1, 30 days prior to scan and Visit 4, 90 days after scan
  Difference in 5-point scale of care partner satisfaction before team care and after amyloid PET scan
Change in care partner assessment of the quality of evaluation after amyloid PET | Visit 1, 30 days prior to scan and Visit 4, 90 days after scan
  Difference in 5-point scale of care partner quality before team care and after amyloid PET scan
Proportion of care partners finding amyloid PET scan worthwhile | Visit 4, 90 days after scan
  Proportion of care partners indicating they would agree to do an amyloid PET again on a yes/no/don't know scale
Proportion exhibiting increased behavior disturbance during amyloid scan visit | Visit 1, Visit 2, Visit 3, and Visit 4 90 days post scan
  % of patients showing a difference in the 44-point Catastrophic Reaction Scale between the median value in all non-scan visits and the value in the amyloid PET scan visit
Percentage of change exhibiting increased behavior disturbance when the diagnosis is given | Visit 1, Visit 3, 60 days
  % of patients showing a difference in the 44-point Catastrophic Reaction Scale between Visit 1 and Visit 3 when learning the result of the scan
Care partner's sustained confidence in diagnosis received after amyloid PET scan | Visit 4, Visit 5, and Visit 6, 270 days post scan
  Care partner confidence in diagnosis received after amyloid PET scan on a 5-point scale
Care partner's sustained confidence in ability to adhere to management plan received after amyloid PET scan | Visit 4, Visit 5, and Visit 6, 270 days post scan
  Care partner confidence in ability to follow management plan outlined by physician after amyloid PET scan on a 5-point scale
Percentage of recommended care practices adhered to after amyloid PET scan | Visit 4, Visit 5, and Visit 6, 270 days post scan
  % of care practices recommended after amyloid PET scan reported by care partner
Percentage of recommended drug management adhered to after amyloid PET scan | Visit 4, Visit 5, and Visit 6, 270 days post scan
  % of drug management options recommended after amyloid PET scan reported by care partner

OTHER OUTCOMES:
Change in the interpretation of amyloid PET scans with semi-quantitative image analysis | within 30 days post amyloid PET scan
  Difference in a 5-point measure of amyloid scan positivity between a qualitative and semi-quantitative image analysis

CONTACTS AND LOCATIONS:
Overall Officials: Norman L. Foster, M.D., Principal Investigator — Director: Center for Alzheimer's Care, Imaging & Research; Chief: Division of Cognitive Neurology; Senior Investigator: The Brain Institute; Professor: Dept. of Neurology University of Utah School of Medicine
Locations (1):
- Center for Alzheimer's Care, Imaging & Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
only de-identified data will be shared

REFERENCES:
- [Background] Naylor MD, Karlawish JH, Arnold SE, Khachaturian AS, Khachaturian ZS, Lee VM, Baumgart M, Banerjee S, Beck C, Blennow K, Brookmeyer R, Brunden KR, Buckwalter KC, Comer M, Covinsky K, Feinberg LF, Frisoni G, Green C, Guimaraes RM, Gwyther LP, Hefti FF, Hutton M, Kawas C, Kent DM, Kuller L, Langa KM, Mahley RW, Maslow K, Masters CL, Meier DE, Neumann PJ, Paul SM, Petersen RC, Sager MA, Sano M, Schenk D, Soares H, Sperling RA, Stahl SM, van Deerlin V, Stern Y, Weir D, Wolk DA, Trojanowski JQ. Advancing Alzheimer's disease diagnosis, treatment, and care: recommendations from the Ware Invitational Summit. Alzheimers Dement. 2012 Sep;8(5):445-52. doi: 10.1016/j.jalz.2012.08.001. PMID 22959699
- [Background] Albert MS, Blacker D. Mild cognitive impairment and dementia. Annu Rev Clin Psychol. 2006;2:379-88. doi: 10.1146/annurev.clinpsy.1.102803.144039. PMID 17716075
- [Background] Mitchell AJ. The clinical significance of subjective memory complaints in the diagnosis of mild cognitive impairment and dementia: a meta-analysis. Int J Geriatr Psychiatry. 2008 Nov;23(11):1191-202. doi: 10.1002/gps.2053. PMID 18500688
- [Background] Matsuda T, Takayama T, Tashiro M, Nakamura Y, Ohashi Y, Shimozuma K. Mild cognitive impairment after adjuvant chemotherapy in breast cancer patients--evaluation of appropriate research design and methodology to measure symptoms. Breast Cancer. 2005;12(4):279-87. doi: 10.2325/jbcs.12.279. PMID 16286908
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Braak H, Braak E. Diagnostic criteria for neuropathologic assessment of Alzheimer's disease. Neurobiol Aging. 1997 Jul-Aug;18(4 Suppl):S85-8. doi: 10.1016/s0197-4580(97)00062-6. PMID 9330992
- [Background] Selkoe DJ. Physiological production of the beta-amyloid protein and the mechanism of Alzheimer's disease. Trends Neurosci. 1993 Oct;16(10):403-9. doi: 10.1016/0166-2236(93)90008-a. PMID 7504355
- [Background] Naslund J, Haroutunian V, Mohs R, Davis KL, Davies P, Greengard P, Buxbaum JD. Correlation between elevated levels of amyloid beta-peptide in the brain and cognitive decline. JAMA. 2000 Mar 22-29;283(12):1571-7. doi: 10.1001/jama.283.12.1571. PMID 10735393
- [Background] Arendash GW, Gordon MN, Diamond DM, Austin LA, Hatcher JM, Jantzen P, DiCarlo G, Wilcock D, Morgan D. Behavioral assessment of Alzheimer's transgenic mice following long-term Abeta vaccination: task specificity and correlations between Abeta deposition and spatial memory. DNA Cell Biol. 2001 Nov;20(11):737-44. doi: 10.1089/10445490152717604. PMID 11788052
- [Background] Mosconi L, McHugh PF. FDG- and amyloid-PET in Alzheimer's disease: is the whole greater than the sum of the parts? Q J Nucl Med Mol Imaging. 2011 Jun;55(3):250-64. PMID 21532539
- [Background] Okello A, Koivunen J, Edison P, Archer HA, Turkheimer FE, Nagren K, Bullock R, Walker Z, Kennedy A, Fox NC, Rossor MN, Rinne JO, Brooks DJ. Conversion of amyloid positive and negative MCI to AD over 3 years: an 11C-PIB PET study. Neurology. 2009 Sep 8;73(10):754-60. doi: 10.1212/WNL.0b013e3181b23564. Epub 2009 Jul 8. PMID 19587325
- [Background] Resnick SM, Sojkova J, Zhou Y, An Y, Ye W, Holt DP, Dannals RF, Mathis CA, Klunk WE, Ferrucci L, Kraut MA, Wong DF. Longitudinal cognitive decline is associated with fibrillar amyloid-beta measured by [11C]PiB. Neurology. 2010 Mar 9;74(10):807-15. doi: 10.1212/WNL.0b013e3181d3e3e9. Epub 2010 Feb 10. PMID 20147655
- [Background] Wolk DA, Price JC, Saxton JA, Snitz BE, James JA, Lopez OL, Aizenstein HJ, Cohen AD, Weissfeld LA, Mathis CA, Klunk WE, De-Kosky ST. Amyloid imaging in mild cognitive impairment subtypes. Ann Neurol. 2009 May;65(5):557-68. doi: 10.1002/ana.21598. PMID 19475670
- [Background] Jack CR Jr, Knopman DS, Jagust WJ, Shaw LM, Aisen PS, Weiner MW, Petersen RC, Trojanowski JQ. Hypothetical model of dynamic biomarkers of the Alzheimer's pathological cascade. Lancet Neurol. 2010 Jan;9(1):119-28. doi: 10.1016/S1474-4422(09)70299-6. PMID 20083042
- [Background] Rowe CC, Villemagne VL. Amyloid imaging with PET in early Alzheimer disease diagnosis. Med Clin North Am. 2013 May;97(3):377-98. doi: 10.1016/j.mcna.2012.12.017. PMID 23642577
- [Background] Thal LJ, Kantarci K, Reiman EM, Klunk WE, Weiner MW, Zetterberg H, Galasko D, Pratico D, Griffin S, Schenk D, Siemers E. The role of biomarkers in clinical trials for Alzheimer disease. Alzheimer Dis Assoc Disord. 2006 Jan-Mar;20(1):6-15. doi: 10.1097/01.wad.0000191420.61260.a8. PMID 16493230
- [Background] Nichols L, Pike VW, Cai L, Innis RB. Imaging and in vivo quantitation of beta-amyloid: an exemplary biomarker for Alzheimer's disease? Biol Psychiatry. 2006 May 15;59(10):940-7. doi: 10.1016/j.biopsych.2005.12.004. Epub 2006 Feb 17. PMID 16487944
- [Background] Yankner BA, Dawes LR, Fisher S, Villa-Komaroff L, Oster-Granite ML, Neve RL. Neurotoxicity of a fragment of the amyloid precursor associated with Alzheimer's disease. Science. 1989 Jul 28;245(4916):417-20. doi: 10.1126/science.2474201.
- [Background] Small GW, Kepe V, Ercoli LM, Siddarth P, Bookheimer SY, Miller KJ, Lavretsky H, Burggren AC, Cole GM, Vinters HV, Thompson PM, Huang SC, Satyamurthy N, Phelps ME, Barrio JR. PET of brain amyloid and tau in mild cognitive impairment. N Engl J Med. 2006 Dec 21;355(25):2652-63. doi: 10.1056/NEJMoa054625. PMID 17182990
- [Background] Mathis CA, Wang Y, Holt DP, Huang GF, Debnath ML, Klunk WE. Synthesis and evaluation of 11C-labeled 6-substituted 2-arylbenzothiazoles as amyloid imaging agents. J Med Chem. 2003 Jun 19;46(13):2740-54. doi: 10.1021/jm030026b. PMID 12801237
- [Background] Verhoeff NP, Wilson AA, Takeshita S, Trop L, Hussey D, Singh K, Kung HF, Kung MP, Houle S. In-vivo imaging of Alzheimer disease beta-amyloid with [11C]SB-13 PET. Am J Geriatr Psychiatry. 2004 Nov-Dec;12(6):584-95. doi: 10.1176/appi.ajgp.12.6.584. PMID 15545326
- [Background] Price JC, Klunk WE, Lopresti BJ, Lu X, Hoge JA, Ziolko SK, Holt DP, Meltzer CC, DeKosky ST, Mathis CA. Kinetic modeling of amyloid binding in humans using PET imaging and Pittsburgh Compound-B. J Cereb Blood Flow Metab. 2005 Nov;25(11):1528-47. doi: 10.1038/sj.jcbfm.9600146. PMID 15944649
- [Background] Mintun MA. Utilizing advanced imaging and surrogate markers across the spectrum of Alzheimer's disease. CNS Spectr. 2005 Nov;10(11 Suppl 18):13-6. doi: 10.1017/s1092852900014188. PMID 16273025
- [Background] Rabinovici GD, Furst AJ, O'Neil JP, Racine CA, Mormino EC, Baker SL, Chetty S, Patel P, Pagliaro TA, Klunk WE, Mathis CA, Rosen HJ, Miller BL, Jagust WJ. 11C-PIB PET imaging in Alzheimer disease and frontotemporal lobar degeneration. Neurology. 2007 Apr 10;68(15):1205-12. doi: 10.1212/01.wnl.0000259035.98480.ed. PMID 17420404
- [Background] Koole M, Lewis DM, Buckley C, Nelissen N, Vandenbulcke M, Brooks DJ, Vandenberghe R, Van Laere K. Whole-body biodistribution and radiation dosimetry of 18F-GE067: a radioligand for in vivo brain amyloid imaging. J Nucl Med. 2009 May;50(5):818-22. doi: 10.2967/jnumed.108.060756. Epub 2009 Apr 16. PMID 19372469
- [Background] Nelissen N, Van Laere K, Thurfjell L, Owenius R, Vandenbulcke M, Koole M, Bormans G, Brooks DJ, Vandenberghe R. Phase 1 study of the Pittsburgh compound B derivative 18F-flutemetamol in healthy volunteers and patients with probable Alzheimer disease. J Nucl Med. 2009 Aug;50(8):1251-9. doi: 10.2967/jnumed.109.063305. Epub 2009 Jul 17. PMID 19617318
- [Background] Vandenberghe R, Van Laere K, Ivanoiu A, Salmon E, Bastin C, Triau E, Hasselbalch S, Law I, Andersen A, Korner A, Minthon L, Garraux G, Nelissen N, Bormans G, Buckley C, Owenius R, Thurfjell L, Farrar G, Brooks DJ. 18F-flutemetamol amyloid imaging in Alzheimer disease and mild cognitive impairment: a phase 2 trial. Ann Neurol. 2010 Sep;68(3):319-29. doi: 10.1002/ana.22068. PMID 20687209
- [Background] Wolk DA, Grachev ID, Buckley C, Kazi H, Grady MS, Trojanowski JQ, Hamilton RH, Sherwin P, McLain R, Arnold SE. Association between in vivo fluorine 18-labeled flutemetamol amyloid positron emission tomography imaging and in vivo cerebral cortical histopathology. Arch Neurol. 2011 Nov;68(11):1398-403. doi: 10.1001/archneurol.2011.153. Epub 2011 Jul 11. PMID 21747004
- [Background] Rinne JO, Wong DF, Wolk DA, Leinonen V, Arnold SE, Buckley C, Smith A, McLain R, Sherwin PF, Farrar G, Kailajarvi M, Grachev ID. [(18)F]Flutemetamol PET imaging and cortical biopsy histopathology for fibrillar amyloid beta detection in living subjects with normal pressure hydrocephalus: pooled analysis of four studies. Acta Neuropathol. 2012 Dec;124(6):833-45. doi: 10.1007/s00401-012-1051-z. Epub 2012 Oct 10. PMID 23053137
- [Background] Thurfjell L, Lotjonen J, Lundqvist R, Koikkalainen J, Soininen H, Waldemar G, Brooks DJ, Vandenberghe R. Combination of biomarkers: PET [18F]flutemetamol imaging and structural MRI in dementia and mild cognitive impairment. Neurodegener Dis. 2012;10(1-4):246-9. doi: 10.1159/000335381. Epub 2012 Feb 1. PMID 22301718
- [Background] Adamczuk K, De Weer AS, Nelissen N, Chen K, Sleegers K, Bettens K, Van Broeckhoven C, Vandenbulcke M, Thiyyagura P, Dupont P, Van Laere K, Reiman EM, Vandenberghe R. Polymorphism of brain derived neurotrophic factor influences beta amyloid load in cognitively intact apolipoprotein E epsilon4 carriers. Neuroimage Clin. 2013 Apr 11;2:512-20. doi: 10.1016/j.nicl.2013.04.001. eCollection 2013. PMID 24179803
- [Background] Duara R, Loewenstein DA, Shen Q, Barker W, Potter E, Varon D, Heurlin K, Vandenberghe R, Buckley C. Amyloid positron emission tomography with (18)F-flutemetamol and structural magnetic resonance imaging in the classification of mild cognitive impairment and Alzheimer's disease. Alzheimers Dement. 2013 May;9(3):295-301. doi: 10.1016/j.jalz.2012.01.006. Epub 2012 Nov 22. PMID 23178035
- [Background] Duff K, Foster NL, Dennett K, Hammers DB, Zollinger LV, Christian PE, Butterfield RI, Beardmore BE, Wang AY, Morton KA, Hoffman JM. Amyloid deposition and cognition in older adults: the effects of premorbid intellect. Arch Clin Neuropsychol. 2013 Nov;28(7):665-71. doi: 10.1093/arclin/act047. Epub 2013 Jun 30. PMID 23817438
- [Background] Leinonen V, Rinne JO, Virtanen KA, Eskola O, Rummukainen J, Huttunen J, von Und Zu Fraunberg M, Nerg O, Koivisto AM, Rinne J, Jaaskelainen JE, Buckley C, Smith A, Jones PA, Sherwin P, Farrar G, McLain R, Kailajarvi M, Heurling K, Grachev ID. Positron emission tomography with [18F]flutemetamol and [11C]PiB for in vivo detection of cerebral cortical amyloid in normal pressure hydrocephalus patients. Eur J Neurol. 2013 Jul;20(7):1043-52. doi: 10.1111/ene.12102. Epub 2013 Feb 11. PMID 23398333
- [Background] Rinne JO, Frantzen J, Leinonen V, Lonnrot K, Laakso A, Virtanen KA, Solin O, Kotkansalo A, Koivisto A, Sajanti J, Karppinen A, Lehto H, Rummukainen J, Buckley C, Smith A, Jones PA, Sherwin P, Farrar G, McLain R, Kailajarvi M, Grachev ID. Prospective flutemetamol positron emission tomography and histopathology in normal pressure hydrocephalus. Neurodegener Dis. 2014;13(4):237-45. doi: 10.1159/000355256. Epub 2013 Nov 27. PMID 24296542
- [Background] Wong DF, Moghekar AR, Rigamonti D, Brasic JR, Rousset O, Willis W, Buckley C, Smith A, Gok B, Sherwin P, Grachev ID. An in vivo evaluation of cerebral cortical amyloid with [18F]flutemetamol using positron emission tomography compared with parietal biopsy samples in living normal pressure hydrocephalus patients. Mol Imaging Biol. 2013 Apr;15(2):230-7. doi: 10.1007/s11307-012-0583-x. PMID 22878921
- [Background] Hatashita S, Yamasaki H, Suzuki Y, Tanaka K, Wakebe D, Hayakawa H. [18F]Flutemetamol amyloid-beta PET imaging compared with [11C]PIB across the spectrum of Alzheimer's disease. Eur J Nucl Med Mol Imaging. 2014 Feb;41(2):290-300. doi: 10.1007/s00259-013-2564-y. Epub 2013 Oct 2. PMID 24085503
- [Background] Pietrzak RH, Lim YY, Neumeister A, Ames D, Ellis KA, Harrington K, Lautenschlager NT, Restrepo C, Martins RN, Masters CL, Villemagne VL, Rowe CC, Maruff P; Australian Imaging, Biomarkers, and Lifestyle Research Group. Amyloid-beta, anxiety, and cognitive decline in preclinical Alzheimer disease: a multicenter, prospective cohort study. JAMA Psychiatry. 2015 Mar;72(3):284-91. doi: 10.1001/jamapsychiatry.2014.2476. PMID 25629787
- [Background] Senda M, Brooks DJ, Farrar G, Somer EJ, Paterson CL, Sasaki M, McParland BJ. The clinical safety, biodistribution and internal radiation dosimetry of flutemetamol ((1)(8)F) injection in healthy Japanese adult volunteers. Ann Nucl Med. 2015 Aug;29(7):627-35. doi: 10.1007/s12149-015-0986-2. Epub 2015 Jun 5. PMID 26044876
- [Background] Curtis C, Gamez JE, Singh U, Sadowsky CH, Villena T, Sabbagh MN, Beach TG, Duara R, Fleisher AS, Frey KA, Walker Z, Hunjan A, Holmes C, Escovar YM, Vera CX, Agronin ME, Ross J, Bozoki A, Akinola M, Shi J, Vandenberghe R, Ikonomovic MD, Sherwin PF, Grachev ID, Farrar G, Smith AP, Buckley CJ, McLain R, Salloway S. Phase 3 trial of flutemetamol labeled with radioactive fluorine 18 imaging and neuritic plaque density. JAMA Neurol. 2015 Mar;72(3):287-94. doi: 10.1001/jamaneurol.2014.4144. PMID 25622185
- [Background] Kelloff GJ, Hoffman JM, Johnson B, Scher HI, Siegel BA, Cheng EY, Cheson BD, O'shaughnessy J, Guyton KZ, Mankoff DA, Shankar L, Larson SM, Sigman CC, Schilsky RL, Sullivan DC. Progress and promise of FDG-PET imaging for cancer patient management and oncologic drug development. Clin Cancer Res. 2005 Apr 15;11(8):2785-808. doi: 10.1158/1078-0432.CCR-04-2626. PMID 15837727
- [Background] Patlak CS, Blasberg RG, Fenstermacher JD. Graphical evaluation of blood-to-brain transfer constants from multiple-time uptake data. J Cereb Blood Flow Metab. 1983 Mar;3(1):1-7. doi: 10.1038/jcbfm.1983.1. PMID 6822610
- [Background] Patlak CS, Blasberg RG. Graphical evaluation of blood-to-brain transfer constants from multiple-time uptake data. Generalizations. J Cereb Blood Flow Metab. 1985 Dec;5(4):584-90. doi: 10.1038/jcbfm.1985.87. PMID 4055928
- [Background] Mintun MA, Larossa GN, Sheline YI, Dence CS, Lee SY, Mach RH, Klunk WE, Mathis CA, DeKosky ST, Morris JC. [11C]PIB in a nondemented population: potential antecedent marker of Alzheimer disease. Neurology. 2006 Aug 8;67(3):446-52. doi: 10.1212/01.wnl.0000228230.26044.a4. PMID 16894106
- [Background] Vlassenko AG, Mintun MA, Xiong C, Sheline YI, Goate AM, Benzinger TL, Morris JC. Amyloid-beta plaque growth in cognitively normal adults: longitudinal [11C]Pittsburgh compound B data. Ann Neurol. 2011 Nov;70(5):857-61. doi: 10.1002/ana.22608. PMID 22162065
- [Background] Rowe CC, Ellis KA, Rimajova M, Bourgeat P, Pike KE, Jones G, Fripp J, Tochon-Danguy H, Morandeau L, O'Keefe G, Price R, Raniga P, Robins P, Acosta O, Lenzo N, Szoeke C, Salvado O, Head R, Martins R, Masters CL, Ames D, Villemagne VL. Amyloid imaging results from the Australian Imaging, Biomarkers and Lifestyle (AIBL) study of aging. Neurobiol Aging. 2010 Aug;31(8):1275-83. doi: 10.1016/j.neurobiolaging.2010.04.007. Epub 2010 May 15. PMID 20472326
- [Background] Fleisher AS, Chen K, Liu X, Roontiva A, Thiyyagura P, Ayutyanont N, Joshi AD, Clark CM, Mintun MA, Pontecorvo MJ, Doraiswamy PM, Johnson KA, Skovronsky DM, Reiman EM. Using positron emission tomography and florbetapir F18 to image cortical amyloid in patients with mild cognitive impairment or dementia due to Alzheimer disease. Arch Neurol. 2011 Nov;68(11):1404-11. doi: 10.1001/archneurol.2011.150. Epub 2011 Jul 11. PMID 21747008
- [Background] Chetelat G, La Joie R, Villain N, Perrotin A, de La Sayette V, Eustache F, Vandenberghe R. Amyloid imaging in cognitively normal individuals, at-risk populations and preclinical Alzheimer's disease. Neuroimage Clin. 2013 Mar 5;2:356-65. doi: 10.1016/j.nicl.2013.02.006. eCollection 2013. PMID 24179789
- [Background] Lundqvist R, Lilja J, Thomas BA, Lotjonen J, Villemagne VL, Rowe CC, Thurfjell L. Implementation and validation of an adaptive template registration method for 18F-flutemetamol imaging data. J Nucl Med. 2013 Aug;54(8):1472-8. doi: 10.2967/jnumed.112.115006. Epub 2013 Jun 5. PMID 23740104
- [Background] Thal D, Beach TG, Zanette M, Heurling K, Buckley C, Smith A. [18F] Flutemetamol amyloid PET in Symptomatic Alzheimer's Disease (AD) and Pathologically Preclinical AD (P-Read) in Comparison to Non-AD Controls: Impact of Cerebral Amyloid Angiopathy. Alzheimer's & Dementia. 2014;10(4):P130.
- [Background] Rowe CC, Dore V, Bourgeat P, et al. Higher AB Burden in Healthy APOE-E4 Carriers is Associated with Subjective Memory Complaints: Results from the Flutemetamol and PIB AIPL Cohorts. Alzheimer's & Dementia. 2014;10(4):P186-P187.
- [Background] Adamczuk K, Schaeverbeke J, Nelissen N, et al. Comparison between semiquantitative measures and reader concordance of amyloid load based on 18F-flutemetamol versus 11C-PIB in cognitively intact older adults. Alzheimer's & Dementia. 2014;10(4):P143.
- [Background] Leinonen V, Rinne JO, Wong DF, Wolk DA, Trojanowski JQ, Sherwin PF, Smith A, Heurling K, Su M, Grachev ID. Diagnostic effectiveness of quantitative [(1)(8)F]flutemetamol PET imaging for detection of fibrillar amyloid beta using cortical biopsy histopathology as the standard of truth in subjects with idiopathic normal pressure hydrocephalus. Acta Neuropathol Commun. 2014 Apr 22;2:46. doi: 10.1186/2051-5960-2-46. PMID 24755237
- [Background] Heurling K, Miki T, Shimada H, et al. Blinded Visual Evaluation and Quantitative SUVR Threshold Classification of [18F]Flutemetamol PET Images in Japanese SUBJECTS. Alzheimer's & Dementia. 2014;10(4):P15.
- [Background] Wolk DA, Duara R, Sadowsky C. [18F]Flutemetamol Amyloid PET Imaging: Outcome of a Phase III Study in Subjects with Amnestic Mild Cognitive Impairment after a 3-Year Follow-Up. Alzheimer's & Dementia. 2014;4(10):P898.
- [Background] Hanseeuw B, Dricot L, Grandin C, Lhommel R, Quenon L, Ivanoiu A. Regional Brain Metabolism and Cortical Thickness in F18-Flutemetamol Amyloid-Positive Versus-Negative Mild Cognitve Impariment Patients. Alzheimer's & Dementia. 2014;10(4):P167-P168.
- [Background] Schaeverbeke J, Adamczuk K, Bruffaerts R, et al. Comparison of 18F-Flutemetamol Uptake and CSF Measurements in Cognitively Intact Older Individuals. Alzheimer's & Dementia. 2014;4(10):P144.
- [Background] AAPM Report No. 96: The Measurement, Reporting, and Management of Radiation Dose in CT. Report of AAPM Task Group 23 of the Diagnostic Imaging Council CT Committee. College Park, MD: American Association of Physicists in Medicine; 2008.